CLINICAL TRIAL: NCT02316392
Title: Imaging and Understanding BOS in Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-6004
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Bronchiolitis Obliterans Syndrome
Keywords: Helium; MRI; Lung transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies of transplanted and explanted lung tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post transplant subjects: Hyperpolarized Helium-3 MRI. Subjects who have had or are scheduled to have a lung transplant
  Interventions: Drug: Hyperpolarized Helium-3 MRI

INTERVENTIONS:
Drug: Hyperpolarized Helium-3 MRI — Subjects will inhale Hyperpolarized Helium-3 gas during the MRI. This gas enhances images and the data collected will be used to determine if it can be used to detect BOS earlier than current standard of care.
  Other Names: Hp-He3 MRI

SUMMARY:
This study is a prospective, non-randomized, longitudinal, observational study that will recruit about 5 lung transplant patients per year for 3 years.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, longitudinal, observational study that will recruit about 5 lung transplant patients per year for 3 years. We will follow these patients at 6 months and 1 year with Hyperpolarized Helium-3 Magnetic Resonance Imaging and image guided bronchial biopsies to detect early BOS and to better understand BO disease progression. The biopsies will provide future research for rapid determination of cellular and molecular mechanisms that lead to BOS and to facilitate identification and validation of translatable pharmaceutical targets.

ELIGIBILITY:
Inclusion Criteria:

* Lung Transplantation within the last 10 years or being assessed for possible lung transplantation.
* Male or female
* 0 to 25 years of age.

Exclusion Criteria:

* Standard MRI exclusion criteria as set forth by the CCHMC Division of Radiology
* Inability to perform 10 second breath hold for 3He MRI scan
* Bleeding disorders

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who have had or are scheduled for lung transplant
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Analysis of MRI imaging to detect BOS compared to biopsy | 3 years
  Analysis of MRI imaging to detect BOS compared to biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD., Principal Investigator — Cincinnati Children's
Locations (1):
- Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share IPD with other researchers at this time. If this plan changes, no identifiable information will be shared.